CLINICAL TRIAL: NCT06875765
Title: Longitudinal Measurement of Synaptic Loss and Cognitive Decline in the Long-term Course of Parkinson's Disease
Brief Title: Long-term Longitudinal Imaging of Presynaptic Terminals in PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S69680
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; PET; UCB-J; PE2I; Positron Emission Tomography
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Longitudinal study design (total follow up time of 7 years) where longitudinal changes of SV2A PET, PE2I PET and clinical rating scales will be compared between patients with PD and healthy controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parkinson disease patients (Experimental)
  Interventions: Other: 11C-UCB-J PET-CT; Other: 18F-PE2I PET-CT; Diagnostic Test: MRI brain
- Healthy controls (Active Comparator)
  Interventions: Other: 11C-UCB-J PET-CT; Other: 18F-PE2I PET-CT; Diagnostic Test: MRI brain

INTERVENTIONS:
Other: 11C-UCB-J PET-CT — Positron Emission Tomography (PET) of synaptic vesicle protein 2A (SV2A) using the radioligand 11C-UCB-J.
Other: 18F-PE2I PET-CT — Positron Emission Tomography (PET) of dopamine transporter (DAT) using the radioligand 18F-FE-PE2I.
Diagnostic Test: MRI brain — Magnetic resonance imaging of brain volume.

SUMMARY:
AIM: To investigate whether SV2A loss spreads from brainstem to cerebral cortex with progression of Parkinson's disease (PD) and to determine whether longitudinal cortical SV2A loss correlates with cognitive decline in PD.

STUDY DESIGN: The investigators will re-invite participants (both patients with PD and healthy controls) of a previous longitudinal study (NCT04243304, S61477) to undergo evaluation approximately 7 years after the initial baseline study visit (i.e. on average 10 years since the first motor symptoms). All participants will undergo clinical assessment of motor and non-motor symptoms (including cognitive testing), as well as 11C-UCB-J PET-CT (targeting synaptic density marker SV2A), 18F-FE-PE2I PET-CT (targeting DAT) and brain MRI.

ELIGIBILITY:
Inclusion Criteria:

* Participation in study S61477 (NCT04243304)

Exclusion Criteria:

* Neuropsychiatric diseases (unrelated to PD for PD patients)
* Major internal medical diseases
* History of alcohol or drug abuse
* Relevant abnormalities on MR brain
* Contraindications for MR
* Pregnancy or breastfeeding
* Previous participation in other research studies involving ionizing radiation with > 1 mSv over past 12 months.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Cross-sectional SV2A at Year 7 | Data analysis will be done when all subjects have undergone Year 7 evaluation.
  Cross-sectional differences (%) in SV2A signal at Year 7 between Parkinson disease patients and controls.
Cross-sectional correlation between clinical scores and SV2A at Year 7 | Data analysis will be done when all subjects have undergone Year 7 evaluation.
  Cross-sectional correlation between clinical scores and SV2A in Parkinson disease patients at Year 7.
Longitudinal SV2A change between baseline and Year 7 | Data analysis will be done when all subjects have undergone Year 7 evaluation.
  Differences (%) in the rate of SV2A change between baseline and Year 7 between Parkinson disease patients and controls.
Longitudinal correlation between clinical scores and SV2A | Data analysis will be done when all subjects have undergone Year 7 evaluation.
  Correlation between progression of the clinical scores and longitudinal SV2A changes in Parkinson disease patients.

SECONDARY OUTCOMES:
Cross-sectional DAT levels at Year 7 | Data analysis will be done when all subjects have undergone Year 7 evaluation.
  Cross-sectional differences (%) in DAT levels at Year 7 between Parkinson disease patients and controls.
Cross-sectional correlation between clinical scores and DAT levels at Year 7 | Data analysis will be done when all subjects have undergone Year 7 evaluation.
  Cross-sectional correlation between clinical scores and DAT levels in Parkinson disease patients at Year 7.
Longitudinal DAT level change between baseline and Year 7 | Data analysis will be done when all subjects have undergone Year 7 evaluation.
  Differences (%) in the rate of DAT level change between baseline and Year 7 between Parkinson disease patients and controls.
Longitudinal correlation between clinical scores and DAT levels | Data analysis will be done when all subjects have undergone Year 7 evaluation.
  Correlation between progression of the clinical scores and longitudinal DAT level changes in Parkinson disease patients.
Longitudinal correlation between SV2A and DAT levels | Data analysis will be done when all subjects have undergone Year 7 evaluation.
  Correlation between SV2A changes and DAT level changes in Parkinson disease patients.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Delva A, Van Weehaeghe D, Koole M, Van Laere K, Vandenberghe W. Loss of Presynaptic Terminal Integrity in the Substantia Nigra in Early Parkinson's Disease. Mov Disord. 2020 Nov;35(11):1977-1986. doi: 10.1002/mds.28216. Epub 2020 Aug 7. PMID 32767618
- [Background] Delva A, Van Laere K, Vandenberghe W. Longitudinal Positron Emission Tomography Imaging of Presynaptic Terminals in Early Parkinson's Disease. Mov Disord. 2022 Sep;37(9):1883-1892. doi: 10.1002/mds.29148. Epub 2022 Jul 12. PMID 35819412